CLINICAL TRIAL: NCT00689442
Title: A 4-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study Evaluating the Safety and Efficacy of JTT-705 600 mg Versus Placebo Administered Once Daily in Combination With Atorvastatin 20 mg in Patients With Low HDL Levels
Brief Title: Safety and Efficacy Study of JTT-705 in Combination With Atorvastatin 20 mg in Patients With Low High-Density Lipoprotein (HDL) Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Shoji Hoshino, DVM, Vice President, Clinical Development, Akros Pharma Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT705-X-03-002
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — dalcetrapib; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): JTT-705 600 mg and atorvastatin 20 mg
  Interventions: Drug: JTT-705 600 mg and atorvastatin 20 mg
- 2 (Placebo Comparator): Placebo and atorvastatin 20 mg
  Interventions: Drug: Placebo and atorvastatin 20 mg

INTERVENTIONS:
Drug: JTT-705 600 mg and atorvastatin 20 mg — * JTT-705 300 mg tablets, 600 mg dose, oral, once daily, immediately following breakfast and/or assessment
  * Atorvastatin 20 mg tablets, 20 mg dose, oral, once daily, immediately following breakfast and/or assessments
  Arms: 1
Drug: Placebo and atorvastatin 20 mg — * Placebo tablet, 2 tablets, oral, once daily, immediately following breakfast and/or assessments
  * Atorvastatin 20 mg tablets, one tablet, oral, once daily, immediately following breakfast and/or assessments
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate safety of JTT-705 and to demonstrate efficacy of JTT-705 compared with placebo when co-administered with atorvastatin 20 mg in patients with low HDL

ELIGIBILITY:
Inclusion Criteria:

* Patients having lipid values as indicated below:
* HDL-C ≤ 1.0 mmol/L (40 mg/dL)
* TG ≤4.5 mmol/L (400 mg/dL)
* Patients with CHD or CHD risk equivalent
* Male and females between 18 and 70 years of age (female patients must be post-menopausal, surgically sterile or using an acceptable form of contraception)

Exclusion Criteria:

* Body Mass Index of ≥ 35 kg/m2
* Females that are pregnant or breast-feeding, and females of child bearing potential who are not using an effective method of contraception
* Concomitant use of medications identified in the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2004-01; Primary Completion 2004-11 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
% change from baseline in HDL-C; inhibition of CETP activity | 4-weeks

SECONDARY OUTCOMES:
% change from baseline in LDL-C and TC/HDL-C | 4-weeks
Plasma concentration of JTT-705 | 4-weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam, Amsterdam, Netherlands